CLINICAL TRIAL: NCT03477877
Title: Indashyikirwa Intervention Trial: Testing a Community-level Programme to Prevent Gender-based Violence in Rwanda
Brief Title: Indashyikirwa IPV Prevention Trial in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council, South Africa (Other)
Collaborators: Department for International Development, United Kingdom (Other Government); CARE Rwanda (Unknown); RWAMREC (Unknown); Laterite (Unknown); London School of Hygiene and Tropical Medicine (Other); Social Development Direct (Unknown); Wellspring Advisors (Unknown); Johns Hopkins University (Other); Rwanda Women's Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC033-10/2015
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Intimate Partner Violence
Keywords: Intimate Partner Violence; Gender-Based violence; Spouse Abuse; Rwanda; Heterosexual Couples; Activists; Opinion Leaders; Social Change; Social-Ecological Model; Diffusion of Innovation; Cluster Randomized Controlled Trial; Community Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: This is a community randomised controlled trial, randomized at the level of sector (Rwandan geographic administrative units are: Province > District > Sector > Cell > Village). 28 sectors spread across 7 districts are participating; randomisation as intervention or control was stratified across districts to ensure adequate geographical spread of program delivery. Within each randomised sector are two separate assessments of impact: (1) A "Couple Cohort" comprised of heterosexual couples who enrol together in a couples training program or similarly situated couples in control communities, surveyed at enrolment, 12 months post-baseline, and 24 months post-baseline. (2) A "Community Survey" designed to measure community diffusion which comprises a repeat cross-sectional population-based household survey of married/cohabiting adults in intervention/control communities who are NOT direct participants in the couples cohort, surveyed at baseline and 24 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indashyikirwa (Experimental): Sectors which receive the full Indashyikirwa programme, including (1) couples training and activist training and support by RWAMREC, and (2) opinion leader training and establishment of women's spaces by the Rwanda Women's Network.
  Interventions: Behavioral: Indashyikirwa Couples Training; Behavioral: Indashyikirwa Activist Training; Behavioral: Indashyikirwa Opinion Leader Training; Other: Indashyikirwa Women's Spaces
- VSLA Only (Active Comparator): Sectors that continue to receive only the village savings and loan association (VSLA) programmes offered by CARE Rwanda
  Interventions: Behavioral: Village Savings and Loan Association (VSLA)

INTERVENTIONS:
Behavioral: Indashyikirwa Couples Training — A training curriculum for heterosexual couples in Rwanda comprising 20 3-hour modules (60 hours total) delivered to groups of 15 couples (30 people). Each module facilitated by male and 1 female facilitator. Curriculum topics include: types and uses of personal and interpersonal power (power within, power over, power with, power to), gender, gender based violence, triggers for intimate partner violence, conflict management, economic development, sexuality, alcohol, social norms and community change. Delivered by RWAMREC.
  Arms: Indashyikirwa
Behavioral: Indashyikirwa Activist Training — This training is offered to a subset of individuals who complete the couples curriculum (randomly selected from among those who are are willing and eligible). These individuals are trained to serve as community activists, teach peers about the types of power (power within, power over, power with, power to), and advocate for community change to prevent intimate partner violence. Delivered by RWAMREC.
  Arms: Indashyikirwa
Behavioral: Indashyikirwa Opinion Leader Training — Training delivered to "opinion leaders" (political office holders, religious leaders, service providers), in intervention communities. Training comprised 8 x 3 hour sessions (24 hours) delivered for groups of up to 40 participants. Introduces Opinion Leaders to the concepts of power (power within, power over, power with, power to) and to essential concepts around women's legal rights. Delivered by Rwanda Women's Network.
  Arms: Indashyikirwa
Other: Indashyikirwa Women's Spaces — Establishment of 1 "Women's Space" per intervention sector -- a physical space with trained facilitators on duty from which support and referrals for women experiencing IPV could be offered and ad hoc programming responsive to community needs and interest can be run. Typical activities include once-off open trainings for community members on the concepts of power (power within, power over, power with, power to), essential concepts around women's legal rights, conflict management in families, etc. Delivered by Rwanda Women's Network.
  Arms: Indashyikirwa
Behavioral: Village Savings and Loan Association (VSLA) — A standard Village Savings and Loan Association program as run nationwide by CARE Rwanda.
  Arms: VSLA Only

SUMMARY:
The purpose of this study is to test whether the Indashyikirwa ("Agents of Change") program is effective at preventing intimate partner violence (IPV) in communities in Rwanda.

Because IPV has many causes, including factors that operate at the individual, couple, and community levels, the Indashyikirwa program is designed with multiple elements targeting multiple levels. A training program for couples covers gender, power, and relationship skills. Individual graduates this program who are interested and eligible go on to an activist training program to help support sustained change in their communities. Parallel activities operate at the Sector level to create and support change at the community level. Sector level activities include (1) training in gender and IPV prevention for local opinion leaders. (2) Establishment of "Women's Spaces," which are drop in centers that provide support and referrals for women experiencing IPV as well as a wide range of community outreach services to educate communities about, gender, power, women's rights, and violence prevention.

Because the intervention is comprised of multiple components and includes elements designed to be delivered at the Sector level, Sectors were chosen as the unit of randomization. 28 sectors spread across 7 districts are participating; randomization as intervention or control was stratified across Districts to ensure adequate geographical spread of program delivery (Rwandan geographic administrative units are: Province > District > Sector > Cell > Village). Within each randomized sector are two separate assessments of program impact: (1) A "Couple Cohort" comprised of heterosexual couples who enrol together in the couples training program (some of whom continue into the activist training) compared to similarly situated couples in control communities who participate only in a standard, ongoing VSLA (village savings and loan association) program. Couples cohort members (both intervention and control) are surveyed at enrolment, 12 months post-baseline, and 24 months post-baseline. (2) A "Community Survey" designed to measure community diffusion of the intervention through the activities of the Women's Spaces, Opinion Leader Trainings, and activities of graduates of the activist training. The community survey comprises a repeat cross-sectional population-based household survey of married/cohabiting adults in intervention communities who are NOT direct participants in any of the formal trainings delivered by intervention implementation partners, conducted at baseline and 24 months only. This survey is designed to look at community level shifts in the occurrence of IPV, as well as changes in support for survivors and changes in attitudes among the general population.

ELIGIBILITY:
Inclusion Criteria:

For the Couples Cohort Study:

1. Member of an active village savings and loan association (VSLA) group or the partner of a VSLA member
2. Between 18 and 49 years old
3. Living with or married to current partner for at least 6 months at baseline
4. Willing and able to give informed consent for participation in research
5. Willing to give contact information of 3 friends, neighbours, or family members who can be used to contact participant over the next 2.5 years
6. Has no current plans to move out of the study area in the next 2.5 years

For the Community Surveys:

1. Resident in the target community for at least 6 months prior to data collection
2. Between 18 and 49 years old
3. Living with or be married to current partner for at least 6 months
4. NOT enrolled in the couples cohort, opinion leader training, or serving as a women's space facilitator (i.e. not otherwise involved in the study)

d. Willing and able to give informed consent for participation in research

Exclusion Criteria (both Couples Cohort and Community Survey):

1. Does not speak Kinyarwanda
2. Unable to provide meaningful informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We did no confirmation of biological sex and accepted all participants as they self-identified.
Enrollment: 8909 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Intimate partner violence with main partner (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of physical or sexual intimate partner violence as assessed by the WHO (World Health Organization) Violence Against Women questions as standardized for the What Works to Prevent Violence Against Women and Girls Programme
Intimate partner violence with main partner (Community Survey) | 24 months
  Experience (for women) or perpetration (for men) of physical or sexual intimate partner violence as assessed by the WHO Violence Against Women questions as standardized for the What Works to Prevent Violence Against Women and Girls Programme
Acceptability of wife beating (Community Survey) | 24 months
  Number of justifications for wife beating endorsed on survey assessment, analyzed separately for male and female participants
Actions to support victims of gender-based violence or combat gender-based violence (Community Survey) | 24 months
  Scores on a checklist of items assessing actions taken to support women who have experienced gender-based violence and/or combat gender-based violence in the community

SECONDARY OUTCOMES:
Newly occuring intimate partner violence with main partner (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of any physical and/or sexual in main intimate partnership during the 12 months before the assessment among participants who DID NOT report physical and/or sexual IPV at baseline
Recurrent physical and/or sexual intimate partner violence (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of any physical and/or sexual in main intimate partnership during the 12 months before the assessment among participants who DID report physical and/or sexual IPV at baseline
Physical intimate partner violence, main partnership (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of any physical violence in main intimate partnership during the 12 months before the assessment
Forced or coerced sex with main partner (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of any forced or coerced sex in main intimate partnership during the 12 months before the assessment
Economic abuse with main partner (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of economic abuse in main intimate partnership during the 12 months before the assessment
Emotional aggression with main partner (Couples Cohort) | 24 months
  Experience (for women) or perpetration (for men) of emotional aggression in main intimate partnership during the 12 months before the assessment
Acceptability of wife beating (Couples cohort) | 24 months
  Number of justifications for wife beating endorsed on survey assessment, analyzed separately for male and female participants
Level of conflict in intimate partnership (Couples Cohort) | 24 months
  Reported sources and frequencies of quarrels with main partner in the past 12 months
Quality of conflict management strategies (Couples Cohort) | 24 months
  Quality of conflict management strategies used in the past 12 months in main intimate partnership (reduced use of negative strategies and increased use of positive strategies)
Couple communication (Couples Cohort) | 24 months
  Frequency of discussing important relationship topics with main partner (her day, his day, her worries or feelings, his worries or feelings, the sexual relationship) in last 4 weeks
Perception of trust, care, and respect in relationship with main partner (Couples Cohort) | 24 months
  Self-reported experience of trust, care, and respect with main partner
Depressive symptoms (Couples Cohort) | 24 months
  Level of depressive symptoms in past week using Center for Epidemiologic Studies Depression Scale (CES-D) short form
Children in household witnessing IPV (Couples Cohort) | 24 months
  Frequency of children witnessing mother being beaten in the past 12 months, per parental report
Problematic alcohol use (Couples Cohort, Men Only) | 24 months
  Measured using AUDIT (Alcohol Use Disorder Identification Test) short form
Help seeking among survivors of IPV (Couples Cohort, Women Only) | 24 months
  Help seeking in past 12 months among women in couples cohort who report experience of physical and/or sexual IPV in the past 12 months
Advising neighbors on relationships (Couples Cohort) | 24 months
  Offering direct support or advice to neighbors regarding IPV or relationship conflict comparing participants who received both couples training and activist training, couples training only, and control participants
Participating in action to prevent IPV (Participants in couples cohort who have received activist training, only) | 24 months
  In past 12 months, participated in a meeting, march, rally or gathering aiming to raise awareness and mobilize people around the issue of family violence comparing participants who received both couples training and activist training, couples training only, and control participants
Self-efficacy for community engagement (Couples Cohort, Women only ) | 24 months
  Confidence to speak at community meetings / to speak at community meetings if people disagree among comparing women who received both couples training and activist training, couples training only, and control participants
Sources of information on IPV and number of times heard (Community Survey) | 24 months
  Frequency of encountering IPV prevention messages in the community
Help seeking among survivors of IPV (Community Survey, women only) | 24 months
  Help seeking in past 12 months among women in community survey who report experience of physical and/or sexual IPV in the past 12 months

OTHER OUTCOMES:
Household earnings (Couples Cohort) | 24 months
  Reported household level earnings in past month
Household debt payments (Couples Cohort) | 24 months
  Reported household debt payments in past month
Food security (Couples Cohort) | 24 months
  Score on standard 2 item assessment of food security
Support physical punishment of children (Couples Cohort) | 24 months
  Endorses statements supporting corporal punishment
Self-rated health (Couples Cohort) | 24 months
  Standard single item assessment
Problematic alcohol use (Couples Cohort, Women only) | 24 months
  Measured using AUDIT (Alcohol Use Disorder Identification Test) short form
PTSD symptoms(Couples Cohort) | 24 months
  Self reports some symptoms indicative of PTSD
Physical intimate partner violence, main partnership (Community Survey) | 24 months
  Experience (for women) or perpetration (for men) of any physical violence in main intimate partnership during the 12 months before the assessment
Forced or coerced sex with main partner (Community Survey) | 24 months
  Experience (for women) or perpetration (for men) of any forced or coerced sex in main intimate partnership during the 12 months before the assessment
Economic abuse with main partner (Community Survey) | 24 months
  Experience (for women) or perpetration (for men) of economic abuse in main intimate partnership during the 12 months before the assessment
Emotional aggression with main partner (Community Survey) | 24 months
  Experience (for women) or perpetration (for men) of emotional aggression in main intimate partnership during the 12 months before the assessment
Children in household witnessing IPV (Community Survey) | 24 months
  Frequency of children witnessing mother being beaten in the past 12 months, per parental report
Support for women working outside the home (Community Survey) | 24 months
  Endorses items supportive of women working outside the home
Change in strategies used to address IPV (Community Survey, women only) | 24 months
  Changes in frequency of checklist of possible strategies for addressing IPV

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Dunkle, PhD, Principal Investigator — Medical Research Council, South Africa; Lori Heise, PhD, Principal Investigator — Johns Hopkins University; Erin Stern, PhD, Principal Investigator — The London School of Hygiene & Tropical Medicine; Lyndsay McLean, PhD, Principal Investigator — Social Development Direct

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dunkle K, Stern E, Chatterji S, Heise L. Effective prevention of intimate partner violence through couples training: a randomised controlled trial of Indashyikirwa in Rwanda. BMJ Glob Health. 2020 Dec;5(12):e002439. doi: 10.1136/bmjgh-2020-002439. PMID 33355268
- [Derived] Gibbs A, Dunkle K, Mhlongo S, Chirwa E, Hatcher A, Christofides NJ, Jewkes R. Which men change in intimate partner violence prevention interventions? A trajectory analysis in Rwanda and South Africa. BMJ Glob Health. 2020 May;5(5):e002199. doi: 10.1136/bmjgh-2019-002199. PMID 32424011
- [Derived] Chatterji S, Stern E, Dunkle K, Heise L. Community activism as a strategy to reduce intimate partner violence (IPV) in rural Rwanda: Results of a community randomised trial. J Glob Health. 2020 Jun;10(1):010406. doi: 10.7189/jogh.10.010406. PMID 32257154